CLINICAL TRIAL: NCT00858832
Title: Reduction of Endometritis After Cesarean Section With the Routine Use of Methergine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 106202
Record Dates: First submitted 2009-03-09; First posted 2009-03-10 (Estimated); Results first posted 2012-09-19 (Estimated); Last update posted 2012-09-19 (Estimated); Status verified 2012-09

CONDITIONS: Endometritis
MeSH Terms: conditions — Endometritis | interventions — Methylergonovine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Methergine (Experimental): Methergine group received Methergine 0.2mg po every 6 hours for two days, plus routine postpartum care.
  Interventions: Drug: Methergine
- No treatment (No Intervention): No treatment group received only routine postpartum care.

INTERVENTIONS:
Drug: Methergine — Scheduled methergine 0.2 mg PO every 6hrs for duration of postpartum stay
  Arms: Methergine

SUMMARY:
Endomyometritis is an "infection in the uterus". It can occur in up to 1 out of 5 women having unplanned cesarean deliveries. Antibiotics are routinely given at the time of Cesarean delivery, but the infection in the uterus can still occur. When endomyometritis occurs it can prolong the woman's stay in the hospital after birth, slow down her recovery time at home, and increase medical costs. Methergine is a medication that is routinely used to stop uterine hemorrhage (excessive bleeding from the uterus) that sometimes happens after delivery. Methergine works by contracting (tightening) the uterus. These contractions also help the uterus to expel or remove parts of the placenta that increase the chance of developing a uterine infection.

This research study is being done to learn if routine use of Methergine can lower the chances of developing a uterine infection after cesarean delivery. Half of the women in this study will receive Methergine for a few days during their hospitalization after cesarean delivery. The other half of the women will not routinely receive Methergine.

ELIGIBILITY:
Inclusion Criteria:

1. Female singleton gravidas
2. Patients receiving non-elective cesarean deliveries after trial of labor
3. No evidence of chorioamnionitis

Exclusion Criteria:

1. Diagnosis of chorioamnionitis
2. Elective cesarean section
3. Unable to provide informed consent
4. Immunocompromised patients and those on antiretroviral drugs
5. Patients with known infection
6. Hypertension (blood pressure greater than 140/90 x 2, six hours apart), including those with a past history, gestational or Preeclampsia.
7. Allergic to ergot alkaloids. This would include people allergic to migraine medicine.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2008-12; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Teefey, MD, Principal Investigator — Univeristy of South Florida OB/GYN
Locations (1):
- Tampa General Hospital, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began 01dec2008 and was terminated 30apr2010. All recruitment was in a hospital.
Pre-assignment Details: There were no washouts or run-ins. Patients were eligible upon the decision for a Cesarean delivery and then consented and randomized.
Groups:
- Methergine: Participants received Methergine 0.2mg orally every 6 hours for 2 days
- No Treatment: Participants received no intervention (no treatment).
Period: Overall Study
Arm/Group | Methergine | No Treatment
Started | 21 (study terminated early due to enrollment deficiencies) | 23
Completed | 20 | 22
Not Completed | 1 | 1
Not completed — became ineligible: delivered vaginally | 1 | 0
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Methergine | No Methergine | Total
Number analyzed (Participants) | 21 | 23 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 23 | 44
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 23 | 44
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Endometritis Incidence
Description: Number of participants who developed endometritis
Time Frame: One year
Measure: Number; unit: participants
Arm/Group | Methergine | No Methergine
Number analyzed (Participants) | 21 | 23
participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Methergine | No Methergine
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/23
Other Adverse Events (participants affected / at risk) | 0/21 | 1/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Methergine (N=21) | No Methergine (N=23)
elevated blood pressure (Pregnancy, puerperium and perinatal conditions) | 0 | 1 — Adverse event was not believed to be related to treatment.

LIMITATIONS AND CAVEATS:
Early termination due to lack of feasibility in completing project; full analysis was not conducted;

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes